CLINICAL TRIAL: NCT00299897
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled Study of Orally Administered SP01A for 28 Days as Monotherapy Treatment in HIV-Infected Patients With Evidence of Resistance to Currently Available Antiretroviral Therapy
Brief Title: SP01A: The Study of an Oral Entry Inhibitor in Treatment-Experienced HIV Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samaritan Pharmaceuticals, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP01A-111-05
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2006-10-27 (Estimated); Status verified 2006-10

CONDITIONS: HIV Infections; Human Immunodeficiency Virus
Keywords: HIV; AIDS; Treatment Resistance; Treatment Failure; Mutations; GP120; Entry Inhibitors; HAART; antiretroviral; antiviral; ARV; CCR5; CXCR4; receptors; intracellular fluid; lipid rafts; cholesterol; chemokine; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Drug: SP01A

SUMMARY:
This is a 28-day, multi-center, placebo-controlled study designed to look at the dose response, efficacy, and safety of SP01A, given as a pill to be swallowed, in the treatment of HIV-infected subjects.

Samaritan has discovered that SP01A affects cholesterol binding, which is directly implicated in the pathogenesis of HIV. It has also been established that drugs of this nature exert an anti-HIV effect in-vitro. These data suggest that SP01A has the potential to reduce HIV virus replication.

One measurement of an HIV infected person's risk of progressing to AIDS is the number of viral particles of HIV in their blood (called a "viral load"). This study is designed to see if SP01A will lower the amount of HIV in an infected individual's blood. Patients will be assigned by chance to 1 of 4 groups. Neither the patient nor the study doctor or nurse will know which dose of the study drug the patient is taking or if he/she is receiving the placebo (a capsule that looks like the study drug but does not contain any active ingredient).

Study drug administration will continue for 28 days. At the end of the 28-day study, the patient will be offered testing of his/her virus for resistance to approved drugs (genotype).

DETAILED DESCRIPTION:
Currently approved antiretroviral medications target either the HIV viral reverse transcriptase (RT), (Nucleoside Reverse Transcriptase Inhibitors (NRTIs) and Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTIs)) or the viral protease, (Protease Inhibitors (PIs)) or inhibit viral fusion with target cells (Fusion Inhibitors). A regimen using a combination of these agents is considered the standard of care and, when effective, results in suppression of the virus below the detection limits.

However, the long-term use of antiretroviral therapy is sometimes hampered by poor compliance due to pill burden, food restrictions, and major side effects that impact Quality of Life. Furthermore, one of the major reasons for therapy failure is the emergence of resistant virus against one or more of the anti-HIV medications or, to some extent, an entire class of drug (cross resistance).

Enfuvirtide (Fuzeon™) was recently approved as an HIV-1 fusion/entry inhibitor, a new class of treatment that prevents fusion of the HIV-1 virus to the CD4+ cell membrane by preventing the conformational changes required for this fusion. Since the mechanism of action of Enfuvirtide is different from other classes of anti-HIV medication, it is effective in patients who have failed other therapies due to emergence of resistant virus. However, a recent study demonstrated the emergence of resistance to Enfuvirtide due to a mutation in viral gp41.

The rapid rate of mutation of HIV-1 and conferred resistance of the virus to current therapies continues to necessitate a need for additional therapeutic agents. To that end, a hypothesis has been suggested regarding the immuno-modulating and anti-viral effects of SP01A in the treatment of HIV infection.

SP01A may affect cholesterol binding, which is directly implicated in the pathogenesis of HIV. Several observations have also established that inhibitors of cholesterol synthesis inhibit cell fusion formation induced by HIV-l and that drugs extracting cholesterol from the cellular membrane exert an anti-HIV-1 effect in-vitro. Taken together, these data may suggest that procaine hydrochloride and SP01A reduces HIV-1 virus replication by modifying the cholesterol content of the cell membrane, rendering it much more difficult for the virus to enter and infect the cell.

There is an urgent need to develop improved new therapeutic agents. SP01A, which targets different viral or cellular components with a new mechanism of action, is being developed and tested by Samaritan Pharmaceuticals, Inc. as a new anti-viral therapeutic agent.

This multi-center, double-blind, randomized, placebo-controlled study of orally administered SP01A as monotherapy in HIV-infected patients with evidence of resistance to currently available antiretroviral therapy was designed to further evaluate the dose response, efficacy, and safety of SP01A. HIV-positive patients will be evaluated during the pre-study period. Following a 2-week washout period (if required), patients will be randomized into one of four study arms and all arms will initiate the 28-day monotherapy study. The first arm will receive 200 mg of SP01A QID. Arm Two will receive 200 mg bid. The third arm will orally administer 400 mg bid. Finally, the fourth arm will receive placebo twice daily.

During the treatment period, patients will make five scheduled visits to the treatment facility on or about Days 1, 8, 15, 22, and 29. During these visits patients will be monitored for viral load and general health parameters. At the conclusion of the 28-day monotherapy study, patients will have optimized viral testing for further treatment.

On Day 43, patients will make their final visit to the treatment facility for post-study evaluation.

ELIGIBILITY:
Inclusion Criteria:

Prior to the first day of study drug:

1. Patient must be capable of giving informed consent prior to the screening visit.
2. Patient is HIV-positive and has treatment-experienced virologic failure or documented resistance. Treatment-experienced virologic failure is defined as patients meeting the following criteria; (1) previous experience with antiretroviral therapy from at least two of the approved antiretroviral classes (i.e. treatment with a nucleoside reverse transcriptase inhibitor, and/or non-nucleoside reverse transcriptase inhibitor, and/or protease inhibitor) for three to six months; (2) increasing HIV RNA after treatment had previously lowered viral load to low or undetectable levels; (3) increased viremia (HIV RNA > 5,000 copies/mL) in at least two viral load tests, one of which can be the screening viral load test, confirming their failing regimen. A patient that is currently on a stable antiretroviral regimen that is successfully suppressing or maintaining viremia at low detectable levels (HIV RNA < 5,000 copies/mL) is not eligible for entry into the study.
3. Patient has been off all antiviral medications including any unapproved or experimental treatment for at least 2 weeks prior to Study Day-1 (baseline).
4. Patient has not taken any experimental medications for at least 4 weeks prior to Screening.
5. Patient is at least 18 years of age and not older than 60 years of age.
6. Patient is capable of adhering to the protocol.
7. Patient has a CD4+ count >/= 100 copies/mL.
8. Patient has a viral load of > 5000 copies/mL.
9. Patient has a Karnofsky score >/= 60.
10. Female patients that are of childbearing potential; (1) have a negative urine pregnancy test at screening, and agree to use a condom and another form of contraception (dual contraception) from the start of the study; or (2) are incapable of becoming pregnant.

Exclusion Criteria:

Patients are ineligible to participate in the study if ANY of the following criteria are met.

1. Patients with known or suspected allergy to procaine hydrochloride.
2. Patients that must take oral or injectable anticholinesterase inhibitors (alone or in combination) for the treatment of myasthenia gravis or as a reversal agent or antagonist to nondepolarizing muscle relaxants such as curariform drugs. Patients using eye medications for glaucoma are not excluded from the study.
3. Patients with SGOT (AST) baseline value >3 times upper limit.
4. Patients with SGPT (ALT) baseline value >3 times upper limit.
5. Patients with Creatinine >2.0 mg/dl.
6. Patients with Absolute Neutrophil count <1,000 cells/mm3.
7. Patients with Platelets baseline value <75,000 cells/µl.
8. Patients that currently have any active opportunistic infection. Prophylaxis for MAI, CMV, PCP, or Herpes is permitted.
9. Females that are pregnant or breast feeding.
10. Female patients of childbearing age who cannot either use dual contraception or abstain from sexual intercourse during the clinical study.
11. Patients with less than 6 months life expectancy.
12. Patients with active hepatitis (viral or drug induced).
13. Patients with cancer, except peripheral (dermal) Kaposi's sarcoma.
14. Patients on dialysis.
15. Patients that currently have an active alcohol or substance abuse.
16. Patients with any medical, psychological, psychiatric or substance use problem that, in the opinion of the principal investigator, will interfere with the patient's ability to complete the study.
17. A patient that is currently on a stable antiretroviral regimen that is successfully suppressing or maintaining viremia at low detectable levels (HIV RNA < 5,000 copies/mL) is not eligible for entry into the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 2006-03

PRIMARY OUTCOMES:
Within treatment group reduction in viral load (log10) in each SP01A active arm as well as within the placebo arm as measured from DAY-1 (Baseline) to DAY-22, and DAY-29 (Study-End).

SECONDARY OUTCOMES:
Reduction in viral load compared across SP01A active arms measured from DAY-1 (Baseline) to DAY-22 and DAY-29 (Study-End).

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Musni, MD, Study Director — Medical Director, Samaritan Pharmaceuticals
Locations (5):
- United States (5):
  - AIDS Healthcare Foundation, Beverly Hills, California
  - Therafirst Medical Centers, Fort Lauderdale, Florida
  - Infectious Disease of Central Florida, Orlando, Florida
  - Triple O Medical Servcies, West Palm Beach, Florida
  - Anderson Medical Group, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Xu J, Lecanu L, Han Z, Yao Z, Greeson J, Papadopoulos V. Inhibition of adrenal cortical steroid formation by procaine is mediated by reduction of the cAMP-induced 3-hydroxy-3-methylglutaryl-coenzyme A reductase messenger ribonucleic acid levels. J Pharmacol Exp Ther. 2003 Dec;307(3):1148-57. doi: 10.1124/jpet.103.055178. Epub 2003 Oct 14. PMID 14560037